CLINICAL TRIAL: NCT01892566
Title: Using mHealth to Respond Early to Acute Exacerbations of COPD in HIV (mREACH)
Brief Title: Using Mobile Health to Respond Early to Acute Exacerbations of COPD in HIV
Acronym: mReach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HL117349; R34HL117349 (NIH)
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: COPD; COPD Exacerbation
Keywords: HIV; mobile health; spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care for COPD (No Intervention): Usual care for AECOPD in the JHHCC consists of patient-initiated contact with the clinic for change in respiratory symptoms. Participants will be asked to complete a weekly symptom diary assessment which will be returned to the study staff at every 3-month visits. Participants contacting research staff with a worsening in respiratory symptoms will be referred to their assigned clinical providers.
- mHealth Intervention (Experimental): For the mHealth intervention, investigators will use of the eResearch Technology, Inc system (ERT®; Philadelphia, PA) for home-based monitoring of spirometry and respiratory symptoms. In conjunction, wireless sensor-based inhalers will monitor the frequency of rescue inhaler use (Asthmapolis®; Madison, WI). As well, on a daily basis, participants in the early identification group will complete eight respiratory symptom questions from the COPD Assessment Test (CAT). Participants' short acting beta-agonist inhaler use will be monitored by an Asthmapolis Spiroscout Inhaler Tracker. Based on participant responses, flags or electronic notifications can be generated. Based on severity of symptoms and guidelines for recommended care, participants will be instructed to self-manage by optimizing inhaler use (if symptoms are mild) or present for an acute care visit at JHHCC if necessary.
  Interventions: Other: mHealth Intervention

INTERVENTIONS:
Other: mHealth Intervention — See arm description
  Other Names: Home spirometer; Inhaler monitor
  Arms: mHealth Intervention

SUMMARY:
Investigators propose to develop methods to improve early identification of acute exacerbations of COPD (AECOPD) among HIV-infected individuals. Investigators hypothesize that earlier identification of acute exacerbations through in-home monitoring of respiratory symptoms, lung function and medication usage will allow appropriate intervention to reduce the morbidity associated with AECOPD. Therefore, the investigators propose using innovative mobile health (mHealth) applications to Respond Early to Acute exacerbations of COPD in HIV (mREACH). COPD is a co-morbidity of HIV with growing recognition, but remains greatly under-recognized among HIV-infected persons. In this application, among HIV-infected individuals with spirometry-confirmed COPD, investigators will conduct a pilot randomized trial of mHealth monitoring compared to usual care to reduce the symptom and clinical burden of AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Has an established longitudinal care provider in Baltimore, MD
* Confirmed COPD defined as post-bronchodilator FEV1/FVC<0.70
* Stable residence for duration of 6 month intervention

Exclusion Criteria:

* Age < 18 years
* Unable/unwilling to provide informed consent
* Failure to present to randomization visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
composite clinical outcome of any COPD-related ER visit or hospitalization | 6 months
  Investigators will assess both patient-reported and clinical outcomes. Both the usual care and intervention arms will complete a paper version of the CAT on a weekly basis. Investigators will compare symptom-free days and time to symptom resolution after an AECOPD. Investigators will also evaluate the composite clinical outcome of any COPD-related ER visit or hospitalization. Additionally, investigators will determine the feasibility, participant acceptability (defined as retention in the study, daily usage of device), and monitoring intensity needed for future trials. Investigators will also collect preliminary data on the number of contacts made to the participant based on automated flags, response of HIV provider, change to medical regimen for COPD care, hospitalization and clinic visits. Investigators will assess changes in respiratory specific quality of life measures using the St. George's Respiratory Questionnaire each month.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kirk, MD MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ALIVE Clinic, Baltimore, Maryland, United States